CLINICAL TRIAL: NCT05389917
Title: Three-Dimensional Vascular Reconstruction of the Pancreas on Multidetector Computed Tomography Images and Its Impact on Patients Undergoing Pancreaticoduodenectomy - A Prospective Observational Study
Brief Title: Three-Dimensional Vascular Reconstruction of the Pancreas on Multidetector Computed Tomography Images and Its Impact on Patients Undergoing Pancreaticoduodenectomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: IEC/2022/92/MA10
Record Dates: First submitted 2022-05-09; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Pancreaticoduodenectomy
Keywords: Inferior Pancreaticoduodenal artery; Multi detector Computed Tomography
MeSH Terms: interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Consecutive adult patients undergoing pancreaticoduodenectomy: All the consecutive patients who undergo pancreaticoduodenectomy will be recruited into the study after obtaining informed consent
  Interventions: Procedure: Pancreaticoduodenectomy

INTERVENTIONS:
Procedure: Pancreaticoduodenectomy — In Pre Operative phase
  64 Slice MD CT scan will be taken in all patients undergoing PD in pre op period 3D reconstruction of Peripancreatic vascular system using MDCT images Measure longitudinal distance between Root of Left renal vein, origin of IPDA Measure distance between origin of SMA , MCA and the IPDA
  In Intraoperative period
  Distance will be measured using standard disposable ruler from Root of Left renal vein to IPDA after Transection of Pancreas followed by specimen removal and to measure the distance between MCA, SMA and IPDA using standard disposable ruler .

SUMMARY:
Three-Dimensional Vascular Reconstruction of the Pancreas on Multi detector Computed Tomography images and its impact on patients undergoing Pancreatoduodenectomy - A Prospective Observational Study IPDA is difficult to identify in pre op in routine CECT images IPDA is difficult to identify in intra op Identification of those major blood vessels (SMA, MCA, Left Renal vein) that lie around the IPDA and then to measure the distances between these major vessels and the IPDA, helps to determine the location of the IPDA

DETAILED DESCRIPTION:
Pancreaticoduodenectomy (PD) is a complex surgical procedure performed for benign and malignant indications .

Vascular anatomy of the pancreatic head, is important in multiple aspects

* Classical arterial anatomy is observed in 55-79% of cases
* Arterial Variation is observed in around 25-30% of cases
* Relationship of the tumor to the blood vessels determines the resectability of tumor The presence of anatomical variations may increase the risk of complications through
* direct (bleeding due to intraoperative vessel injury)
* indirect (postoperative ischemia of tissues and anastomotic leakage) Preoperative understanding of the vascular anatomy of the pancreatic head is important in order to reduce intraoperative bleeding.
* IPDA is difficult to identify in pre op in routine CECT images. It is identified in only 20% of patients.
* IPDA is difficult to identify in intra op because- It generally originates from the posterior wall of superior mesenteric artery (SMA).The origin of IPDA frequently varies, which makes it difficult to identify in some patients. It is surrounded by dense lymphovascular tissue, which makes it difficult to identify IPDA during surgery.

IPDA can be identified in up to 86% of the time using 3D MDCT . Identification of those major blood vessels (SMA, MCA, Left Renal vein) that lie around the IPDA and then to measure the distances between these major vessels and the IPDA, helps to determine the location of the IPDA.

In the existing studies, they have not defined the impact of identifying IPDA on intra operative parameters ( Operative time, Blood loss) These studies have not used uniform landmarks in the identification of IPDA

ELIGIBILITY:
Inclusion Criteria:

• Consecutive Patients undergoing pancreaticoduodenectomy during the study period at ILBS

Exclusion Criteria:

* If surgery is not proceeded for any cause like Presence of metastasis, Unreconstructable portal or SMV involvement , SMA involvement of >180 degree
* Refusal for consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients undergoing pancreaticoduodenectomy during the study period at ILBS
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-05-30 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Probability of identifying IPDA with in 1 cm of anticipated location from Left renal vein determined by preoperative 3D reconstructed MDCT images. | During the Procedure
  During the procedure distance will be measured between root of Left Renal vein to Origin of IPDA

SECONDARY OUTCOMES:
To correlate the location of IPDA predicted by 3D reconstruction of preoperative MDCT images with actual intraoperative location of MCA and SMA, after specimen removal | During the Procedure
  During the procedure distance will be measured between Origin of SMA and MCA to Origin of IPDA
To correlate the early ligation of IPDA with Blood Loss and Operative time | During the Procedure
  Blood Loss during the procedure and time required to complete the pancreaticoduodenectomy procedure
Spectrum of arterial anomalies encountered during Pancreaticoduodenectomy | During The Procedure
  Anatomy of vascular arcades arising from the celiac and superior mesenteric arteries will be noted during the procedure
To compare operative time between patients who undergo pre operative 3D vascular reconstruction on MD CT followed by Pancreaticoduodenectomy versus historical controls who have undergone pancreaticoduodenectomy at ILBS | During the Procedure
  Operative time of patients who have undergone pancreaticoduodenectomy during the study period is compared with historical cohorts
To compare blood loss between patients who undergo pre operative 3D vascular reconstruction on MD CT followed by Pancreaticoduodenectomy versus historical controls who have undergone pancreaticoduodenectomy at ILBS | During the Procedure
  Blood loss of patients who have undergone pancreaticoduodenectomy during the study period is compared with historical cohorts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tomimaru Y, Tanaka K, Noguchi K, Hatano H, Eguchi H, Dono K. Distance from Left Renal Vein to Inferior Pancreaticoduodenal Artery: A Landmark for Identifying Inferior Pancreaticoduodenal Artery in Pancreatoduodenectomy. Dig Surg. 2017;34(4):335-339. doi: 10.1159/000453553. Epub 2017 Jan 19. PMID 28099958
- [Background] Horiguchi A, Ishihara S, Ito M, Asano Y, Yamamoto T, Miyakawa S. Three-dimensional models of arteries constructed using multidetector-row CT images to perform pancreatoduodenectomy safely following dissection of the inferior pancreaticoduodenal artery. J Hepatobiliary Pancreat Sci. 2010 Jul;17(4):523-6. doi: 10.1007/s00534-009-0261-9. Epub 2010 Feb 9. PMID 20714842
- [Background] Fang CH, Kong D, Wang X, Wang H, Xiang N, Fan Y, Yang J, Zhong SZ. Three-dimensional reconstruction of the peripancreatic vascular system based on computed tomographic angiography images and its clinical application in the surgical management of pancreatic tumors. Pancreas. 2014 Apr;43(3):389-95. doi: 10.1097/MPA.0000000000000035. PMID 24622068
- [Background] Perwaiz A, Singh A, Singh T, Chaudhary A. Incidence and management of arterial anomalies in patients undergoing pancreaticoduodenectomy. JOP. 2010 Jan 8;11(1):25-30. PMID 20065548
- [Background] Sim JS, Choi BI, Han JK, Chung MJ, Chung JW, Park JH, Han MC. Helical CT anatomy of pancreatic arteries. Abdom Imaging. 1996 Nov-Dec;21(6):517-21. doi: 10.1007/s002619900117. PMID 8875875
- [Background] Patel BN, Giacomini C, Jeffrey RB, Willmann JK, Olcott E. Three-dimensional volume-rendered multidetector CT imaging of the posterior inferior pancreaticoduodenal artery: its anatomy and role in diagnosing extrapancreatic perineural invasion. Cancer Imaging. 2013 Dec 30;13(4):580-90. doi: 10.1102/1470-7330.2013.0051. PMID 24434918